CLINICAL TRIAL: NCT07237256
Title: No Chemotherapy in Intermediate-risk HR+ HER2- Early Breast Cancer Treated With Ribociclib (LEE-011) in the Adjuvant Setting, a Non-inferiority Phase III Trial
Brief Title: Chemotherapy De-escalation in HR +, HER2-, Intermediate-risk Early Breast Cancer Treated With Adjuvant Ribociclib
Acronym: NoLEEta
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Novartis (Industry); SOLTI Breast Cancer Research Group (Other); GBG Forschungs GmbH (Other); Latin American Cooperative Oncology Group (Other); Gruppo Italiano Mammella (GIM) (Other); BOOG Study Center (Other); Canadian Cancer Trials Group (Network); Swiss Cancer Institute (Other); Menarini Silicon Biosystems, INC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-BCG-2501; 2025-520979-13-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: De-escalation; Chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Drug Therapy; ribociclib

STUDY DESIGN:
Intervention Model Description: * Investigational arm (Arm A): ribociclib and endocrine therapy (ET)
  * Control arm (Arm B): chemotherapy followed by ribociclib and endocrine therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational arm (Arm A) (Experimental): Ribociclib and endocrine therapy (ET)
  Interventions: Other: De-escalation
- Control arm (Arm B) (Other): Chemotherapy followed by ribociclib and endocrine therapy
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — Control arm
  Other Names: Ribociclib; Adjuvant hormonotherapy
  Arms: Control arm (Arm B)
Other: De-escalation — De-escalation of the chemotherapy in the adjuvant setting
  Other Names: Ribociclib; Adjuvant hormonotherapy
  Arms: Investigational arm (Arm A)

SUMMARY:
The advent of CDK4/6 inhibitors (drugs designed to block the action of CDK4/6 proteins, which play a key role in cell proliferation) has improved treatment prospects for patients with metastatic breast cancer whose tumour cells express hormone receptors but not the HER2 protein (HR+/HER2-). The NATALEE study showed that the addition of ribociclib for three years to conventional adjuvant hormone therapy (i.e. after surgery) prolonged survival free of invasive disease (i.e. extending to surrounding tissues) in patients with early HR breast cancer+ /HER2-. Unlike other studies, NATALEE included a group of patients at intermediate risk of recurrence, usually treated with adjuvant chemotherapy before receiving hormone therapy. However, the benefit of adjuvant chemotherapy in these patients is uncertain. The hypothesis of the NoLEEta study is that by using the CDK 4/6 inhibitor, patients could avoid adjuvant chemotherapy and therefore be spared the side-effects associated with this chemotherapy, without reducing the efficacy of the treatment.

DETAILED DESCRIPTION:
The advent of CDK4/6 inhibitors has changed the outlook of patients with metastatic hormone receptor-positive (HR+) HER2- breast cancer. Moreover, including CDK4/6 inhibitors in the adjuvant treatment regimens strategies has led to significant gains in disease-free survival.

The phase III NATALEE trial demonstrated the efficacy of an adjuvant three-year treatment with ribociclib in prolonging invasive disease-free survival (iDFS) in patients with intermediate and high-risk HR+ HER2- early breast cancer.

Contrarily to similar studies of CDK4/6 inhibitors in this setting, NATALEE included a group of patients with intermediate clinical risk (pT1-2 pN1, pT3-4 pN0 or pT2 pN0 with histological grade 3 or grade 2 with Ki67≥ 20%). These patients are usually considered for adjuvant chemotherapy based on their clinicopathological conditions or the results of a genomic signature (e.g. Oncotype Dx). Nevertheless, the benefit of adjuvant chemotherapy in these patients is uncertain (and likely small) in the context of an adjuvant treatment strategy that includes a CDK 4/6 inhibitor.

As such, a de-escalation trial could demonstrate that patients with intermediate-risk breast cancer treated with CDK4/6 inhibitors could be spared the dreaded chemotherapy side effects while ensuring similar survival outcomes.

In order to be generalizable and practice changing, a trial in this setting should aim to be as pragmatic as possible, particularly in inclusion criteria, with the required resources for patient inclusion and delivery of care being as similar as possible to those employed in usual care. As such, chemotherapy eligibility should be defined similarly to routine clinical practice in the participating centers (i.e. using routine clinicopathological parameters and/or genomic signatures).

While single-arm designs could help address non-inferiority in the previously mentioned setting, they are usually compared to historical controls and lack external validation. Moreover, in some settings, like early breast cancer, the standard of care may change relatively quickly (e.g. Oncotype Dx-based chemotherapy de-escalation or adjuvant CDK4/6 inhibitors use), rendering the comparison to historical controls challenging, limiting the study conclusions and their impact on clinical practice. Finally, there is no consensus on the optimal non-inferiority threshold in single-arm trials using historical controls as a comparator. As such, randomized controlled non-inferiority trials with a strict non-inferiority margin remain the gold standard design to prove that a de-escalated treatment regimen is safe and advantageous, and the only ones capable of producing level IA evidence according to ESMO (Trapani et al., Annals of Oncology 2022).

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have signed a written informed consent prior to any trial-specific screening procedure.

   Note: When the patient is physically unable to give their written consent, an impartial witness of their choice, independent from the investigator or the sponsor, can confirm in writing the patient's consent.
2. Patient is ≥ 18 years old.
3. Patient is female with known menopausal status at the time of randomization.

   Post-menopausal status is defined as:
   1. Patient underwent bilateral oophorectomy, or
   2. Age ≥ 60 years, or
   3. Age < 60 years and either amenorrhea for 12 or more months (in the absence of chemotherapy, tamoxifen, toremifene or ovarian suppression) or Follicle-stimulating hormone (FSH) and plasma estradiol are in the postmenopausal ranges per local normal ranges.
   4. If taking tamoxifen or toremifene and age <60 years, then FSH and plasma estradiol level in postmenopausal ranges.
4. The following criteria must be met for histologically confirmed invasive breast carcinoma, as determined by the local pathologist:

   1. Pathological stage (8th edition of the AJCC), including pT2 pN0 Grade 3 or pT2 pN0 Grade 2 with Ki67≥20% or pT0-2 pN1 or pT3-4 pN0
   2. ER-positive (with tumor cells showing ≥10% ER staining) and HER2-negative according to the most recent ASCO/CAP guidelines.

   Note: Multifocal and multicentric tumors are allowed if they meet the clinical stage II criteria of the 8th Edition of the AJCC. All tumors must be ER-positive and HER2-negative. Patients with bilateral invasive breast cancer (diagnosed simultaneously or within 6 months of each other) are eligible if all lesions tested on both sides are ER+ (ie, ≥10% positive stained cells) and HER2- AND adequate surgery has been performed in both breasts.
5. Chemotherapy eligible per investigator decision, based on clinicopathological findings or the results of any genomic signature.
6. Patient has no contraindication for the adjuvant endocrine therapy (ET) or chemotherapy in the trial and is planned to be treated with ET for 5 years (after randomization date) or more.
7. Curative surgery for the invasive disease must have been performed with negative surgical margins within 12 weeks before randomization. If positive surgical margins, patients are eligible if revision surgery or other adequate local treatment (i.e local radiotherapy) is planned.
8. Women of childbearing potential (CBP) must have a confirmed negative serum pregnancy test (β-hCG) before starting study treatment.
9. Women of childbearing potential must agree to use one effective form of contraception during trial treatment and up to 21 days after the last dose of study drugs or longer, if required per standard of care;
10. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 within 28 days prior to randomization.
11. Adequate hematological, renal, and hepatic function, as outlined below:

    1. Absolute neutrophil count (ANC) ≥1.5 x 10⁹/L
    2. Platelet count ≥100 x 10⁹/L
    3. Hemoglobin ≥9 g/dL
    4. Total bilirubin < ULN. Patients with known Gilbert syndrome may be enrolled with total bilirubin ≤3 x ULN or direct bilirubin ≤1.5 x ULN
    5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <2.5 x ULN
    6. Serum creatinine ≤1.5 mg/dL or calculated creatinine clearance ≥60 mL/min/1.73m² (CKD-EPI equation (2021))
    7. Potassium, total calcium (corrected for serum albumin), and magnesium should be within institutional normal limits or corrected to within normal limits using supplements before the first dose of study medication.
12. Standard 12-lead ECG values assessed, as:

    1. QTcF interval (QT interval using Fridericia's correction) at screening < 450 milliseconds (msec)
    2. Resting heart rate 50-100 beats per minute (determined from the ECG)
13. Patient must be willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other trial procedures.
14. Absence of any psychological, familial or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.
15. Patients must be affiliated to a Social Security System (or equivalent) based on local regulations.

Exclusion Criteria:

1. Patient has received any neoadjuvant chemotherapy since her breast cancer diagnosis or has received any prior CDK4/6 inhibitor.
2. Breast cancer diagnosed while patient was receiving tamoxifen, raloxifene or aromatase inhibitors (AIs) for reduction in risk ("chemoprevention") of breast cancer and/or treatment for osteoporosis within the last 2 years prior to randomization.
3. Patient with a known hypersensitivity to any of the excipients of ribociclib and/or ET (e.g. rare hereditary problems of galactose intolerance, the Lapp lactase deficiency, glucose-galactose malabsorption, and soy or peanut allergy).
4. Patient with evidence or history of distant metastases of breast cancer beyond regional lymph nodes (stage IV according to AJCC 8th edition), inflammatory breast cancer, breast cancer recurrence (local or distant) or a different primary breast cancer.
5. Patient has a concurrent invasive malignancy or a prior invasive malignancy whose treatment was completed within 2 years before randomization. Note: Patients with adequately treated basal or squamous cell skin carcinoma or curatively resected cervical cancer in situ are eligible.
6. Patients whose breast cancer is considered as endocrine therapy insensitive, as determined by investigator's opinion; this may include (but is not limited to) breast cancer classified as " basal like " by molecular signatures (if available in the patient file) and/or breast cancer with persistently high proliferation after pre-operative endocrine therapy.
7. Patient has had major surgery within 14 days prior to study treatment initiation.
8. Patient has known history of human immunodeficiency virus (HIV) infection (testing is not mandatory) whose antiretroviral therapy (ART) has a known strong CYP3A4 inhibitor with potential for DDI with ribociclib. Patients with HIV may be enrolled if they fulfil the criteria recommended by FDA and ASCO guidelines (FDA Guidance, Uldrick et al. 2017):

   1. CD4+ T-cell (CD4+) counts ≥ 350 cells/µL, AND
   2. No history of AIDS-defining opportunistic infections within the past 12 months (prophylactic antimicrobials allowed if no drug-drug interactions or overlapping toxicities), AND
   3. On established ART which is not a strong CYP3A4 inhibitor, for at least 4 weeks and have an HIV viral load less than 400 copies/mL prior to enrolment. Effective ART is defined as a drug, dosage, and schedule associated with reduction and control of the viral load.
9. Patient has known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection (testing is not mandatory).
10. Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality, including any of the following:

    1. History of documented myocardial infarction (MI), angina pectoris, symptomatic pericarditis, or coronary artery bypass graft within 6 months prior to trial entry.
    2. Documented cardiomyopathy.
    3. Left Ventricular Ejection Fraction (LVEF) < 50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO) (testing not mandatory)
    4. Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome, or any of the following:

       * Risk factors for Torsades de Pointes (TdP) including uncorrected hypocalcemia, hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia.
       * Concomitant medication(s) with a known risk to prolong the QT interval and/or known to cause TdP that cannot be discontinued or replaced by safe alternative medication (e.g. within 5 half-lives or 7 days prior to starting trial treatment).
       * Inability to determine the QTcF interval.
    5. Clinically significant cardiac arrhythmias (e.g. ventricular tachycardia), complete left bundle branch block, high-grade Atrioventricular (AV) block (e.g. bifascicular block, Mobitz type II and third degree AV block).
    6. Uncontrolled arterial hypertension with systolic blood pressure >160 mmHg.
11. Presence of any other medical conditions, including respiratory or metabolic dysfunction, physical examination findings, or laboratory results that raise reasonable suspicion of a contraindication to the use of an experimental drug, potential impact on compliance with the study protocol, influence on result interpretation, or increased risk of treatment complications for the patients (such as severe dyspnea at rest or requiring oxygen therapy, history of major surgical resection involving the stomach or small bowel, preexisting Crohn's disease or ulcerative colitis, or a preexisting chronic condition resulting in clinically significant diarrhea).
12. Previous history of pneumonitis, regardless of cause.
13. Patient is currently receiving any of the following substances within 7 days before randomization and which cannot be stopped within seven days prior to the start of treatment:

    1. Concomitant medications, herbal supplements, and/or fruits (e.g. grapefruit, pummelos, starfruit, Seville oranges) and their juices that are known as strong inhibitors or inducers of CYP3A4/5
    2. Medications that have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5
    3. Any medication prohibited according to the instructions for goserelin, leuprolide or triptorelin (pre-menopausal patients), anastrozole, exemestane, letrozole, or ribociclib.
    4. Medications known to have a risk of prolonging the QT interval or causing Torsades de Pointes.
14. Patient is concurrently using hormone replacement therapy. Estrogen replacement therapy discontinued less than two weeks prior to the start of treatment.
15. Patient is currently receiving or has received systemic corticosteroids ≤ 2 weeks prior to starting trial treatment, or has not fully recovered from side effects of such treatment.

    Note: The following uses of corticosteroids are permitted: a short duration (<5 days) of systemic corticosteroids; any duration of topical applications (e.g. for rash), inhaled sprays (e.g. for obstructive airways diseases), eye drops or local injections (e.g. intra-articular).
16. Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the Investigator's judgment, cause unacceptable safety risks, contraindicate patient participation in the clinical trial or compromise compliance with the protocol (e.g. chronic pancreatitis, chronic active hepatitis, liver cirrhosis or any other significant liver disease, active untreated or uncontrolled fungal, bacterial or viral infections, active infection requiring systemic anti-bacterial therapy, etc.) or limit life expectancy to ≤5 years.
17. Participation in other studies involving investigational drug(s) within 30 days prior to randomization or within 5 half-lives of the investigational drug(s) (whichever is longer), or participation in any other type of medical research judged not to be scientifically or medically compatible with this trial. If the patient is enrolled or planned to be enrolled in another study that does not involve an investigational drug, the agreement of the sponsor is required to establish eligibility.
18. Inability or unwillingness to swallow oral pills.
19. Presence of malabsorption syndrome or any other condition that could hinder the absorption of study drugs in the gastrointestinal tract.
20. Any psychological, familial, sociological, or geographical factors that may impede adherence to the study protocol and follow-up schedule.
21. Pregnant or breast-feeding (lactating) women or women who plan to become pregnant or breast-feed during the first 48 months of adjuvant therapy.
22. Persons deprived of their liberty or under protective custody or guardianship.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3902 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2033-11-30 (Estimated); Study Completion 2037-12-31 (Estimated)

PRIMARY OUTCOMES:
Invasive breast cancer-free survival (iBCFS) | From ramdomization to iBCFS, up to 12 years.
  iBCFS is defined as the time from the date of randomization to the date of the first event of invasive ipsilateral breast tumor recurrence, local-regional invasive recurrence, distant recurrence, death (any cause) or invasive contralateral breast cancer as assessed by investigator.

SECONDARY OUTCOMES:
Invasive disease-free survival (iDFS) | From ramdomization to iDFS event, up to 12 years.
  iDFS is defined as the time from date of randomization to the date of the first iDFS event that is: i) same event as IBCFS, or ii) secondary invasive non breast cancer.
Distance disease-free survival (DDFS) | From ramdomization to DDFS event, up to 12 years.
  DDFS is defined as the time from the date of randomization to the date of the first event of distant recurrence, death (any cause), or second primary non-breast invasive cancer (excluding basal and squamous cell carcinomas of the skin).
Overall survival (OS) | From ramdomization to death from any cause, up to 12 years.
  OS is defined as the time from the date of randomization to the date of death due to any cause
Type of iBCFS event | From ramdomization to iBCFS event, up to 12 years.
  To evaluate the rate of the different types of iBCFS events in each treatment arm
Acute and late toxicity during the study focusing on grade ≥2 | Throughout study completion, up to 8.5 years.
  The National Cancer Institute-Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5) is widely accepted in the community of oncology research as the leading rating scale for adverse events. This scale, divided into 5 grades (1 = "mild", 2 = "moderate", 3
  = "severe", 4 = "life-threatening", and 5 = "death")
Quality of life questionnaire - Core 30 (QLQ-C30) | At baseline, 3 months, 6 months, 1 year, 2 years, 3 years, 5 years, 8.5 years from randomization.
  Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials. The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of Life Questionnaire - Breast cancer module (QLQ-BR42) | At baseline, 3 months, 6 months, 1 year, 2 years, 3 years, 5 years, 8.5 years from randomization.
  This EORTC breast cancer specific questionnaire is intended to supplement the QLQ-C30.
  The QLQ-BR42 incorporates nine multi-item scales to assess body image, sexual functioning, breast satisfaction, systemic therapy side effects, arm symptoms, breast symptoms, endocrine therapy symptoms, skin mucosis symptoms, endocrine sexual symptoms. In addition, single items assess sexual enjoyment, future perspective and being upset by hair loss. All items are rated on a four-point Likert-type scale (1 = "not at all", 2 = "a little", 3 = "quite a bit", and 4 = "very much"), and are linearly transformed to a 0-100 scale. Higher scores indicate more severe symptoms or problems for all items.

CONTACTS AND LOCATIONS:
Overall Officials: François-Clément BIDARD, PhD, Principal Investigator — Institut Curie
Locations (39):
- France (39):
  - Clinique de l'Europe, Amiens
  - Institut de Cancérologie de l'Ouest - Site Paul Papin, Angers
  - Centre Hospitalier d'Auxerre, Auxerre
  - Centre Hospitalier Universitaire de Besancon, Besançon
  - Institut Bergonié, Bordeaux
  - Centre Francois Baclesse, Caen
  - CH William Morey, Chalon-sur-Saône
  - Centre Hospitalier Métropole de Savoie, Chambéry
  - Centre Hospitalier de Cholet, Cholet
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges François Leclerc, Dijon
  - CHI Fréjus St-Raphaël, Fréjus
  - Centre Hospitalier Départemental de Vendée, La Roche-sur-Yon
  - Clinique Victor Hugo, Le Mans
  - Centre Hospitalier le Mans, Le Mans
  - Centre Hospitalier Universitaire de Limoges, Limoges
  - Centre Leon Berard, Lyon
  - Hôpital privé Jean Mermoz, Lyon
  - Institut Paoli Calmettes, Marseille
  - Centre Hospitalier ANNECY GENEVOIS, Metz-Tessy
  - Centre de Cancerologie du Grand Montpellier, Montpellier
  - Hopital Privé du Confluent, Nantes
  - Centre Antoine Lacassagne, Nice
  - Hopital Diaconesses-Croix Saint Simon, Paris
  - Centre Hospitalier de Pau, Pau
  - CARIO - Centre Armoricain Radiothérapie Imagerie Médicale et Oncologie, Plérin
  - Clinique de la Croix du Sud, Quint-Fonsegrives
  - Institut Jean Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut Curie - Hôpital René Huguenin, Saint-Cloud
  - Institut de Cancérologie de l'Ouest - Site René Gauducheau, Saint-Herblain
  - Clinique Mutualiste de l'Estuaire, Saint-Nazaire
  - Centre Paul Stauss, Strasbourg
  - Hôpitaux du Léman, Thonon-les-Bains
  - Institut Claudius Regaud, Toulouse
  - Centre Hospitalier de Tours - Hopital Bretonneau, Tours
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients.